CLINICAL TRIAL: NCT05555875
Title: A Clinical Trial Aimed at Evaluating Factors Contributing to Patient Engagement With Digital Mental Health Interventions
Brief Title: Toward Understanding Drivers of Patient Engagement With Digital Mental Health Interventions - Part II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica M. Lipschitz, Ph.D., Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P001673; K23MH120324 (NIH)
Record Dates: First submitted 2022-08-22; First posted 2022-09-27 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Depression; Anxiety Disorders
Keywords: Mobile app; Engagement; Depression; Anxiety; Micro-randomized trial
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 2x2 factorial trial with micro-randomization in automated motivational messaging arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IntelliCare with Automated Motivational Messaging and Coach Support (Experimental): IntelliCare Plus mobile application intervention with two engagement strategies, automated motivational messaging and coach support.
  Interventions: Behavioral: IntelliCare Plus
- IntelliCare with Automated Motivational Messaging (Experimental): IntelliCare Plus mobile application intervention with one engagement strategy, automated motivational messaging.
  Interventions: Behavioral: IntelliCare Plus
- IntelliCare with Coach Support (Experimental): IntelliCare Plus mobile application intervention with one engagement strategy, coach support.
  Interventions: Behavioral: IntelliCare Plus
- IntelliCare Alone (Active Comparator): IntelliCare Plus mobile application intervention with no additional engagement strategy applied.
  Interventions: Behavioral: IntelliCare Plus

INTERVENTIONS:
Behavioral: IntelliCare Plus — Mobile-app-based digital mental health intervention for individuals struggling with depression and/or anxiety. The app reflects components of evidence-based psychological treatments such as cognitive-behavioral therapy.

SUMMARY:
This study is a clinical trial that evaluates what drives patient engagement and tests the impact of two strategies-automated motivational push messaging and coach support-to improve engagement with an evidence-based mobile app intervention for depression and/or anxiety.

DETAILED DESCRIPTION:
This 8-week, clinical trial involves primary care patients with clinically significant depression and/or anxiety recruited via provider referral. Participants will received access to a digital mental health intervention with known efficacy and be randomized to an engagement strategy condition--a previously-validated Coach Support protocol (CS), a newly-developed automated motivational messaging protocol (AMM), both or neither. To further understand how messages in the AMM arms function, message delivery will be micro-randomized: each day participants will be randomized to receive a message or not, such that they receive an average of 4.2 messages/week. Micro-randomization allows causal inference about the near-term impact of message delivery (i.e., are AMMs a cue to action) and the relationship between message impact and context (e.g., day in study). Measured outcome data will include level of engagement (operationalized as minutes of intervention use) and weekly self-reports of clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Mass General Brigham primary care patient
* Age 18-75
* Clinically significant symptoms of depression (Patient Health Questionnaire-9 (PHQ-9) greater than or equal to 10) and/or anxiety (Generalized Anxiety Disorder-7 (GAD-7) greater than or equal to 8)
* Owns a smartphone capable of running the study applications
* Fluent in English.

Exclusion Criteria:

* Diagnosis of bipolar I or bipolar II disorder per patient report or the patient's medical record
* Diagnosis of any psychotic disorder per patient report or the patient's medical record
* Current substance use disorder per patient report or the patient's medical record
* Acute and/or unstable medical problem that may interfere with participation (e.g., scheduled for surgery in the next two months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Minutes of Intervention Use - Distal (Long-Term) | 8-week intervention period
  Intervention use logs will be collected continuously and automatically throughout the intervention period on the system backend. Intervention engagement will be operationalized as minutes of active use over the intervention period.
Intervention Engagement Within 3 Hours Following a Decision Point - Proximal (Short-Term) | For 3 hours after each decision point, over the 8-week intervention period
  Intervention use logs will be collected continuously and automatically throughout the intervention period on the system backend. Proximal Intervention engagement will be operationalized as whether or not the intervention was used within 3 hours of a decision point (i.e., the point at which participants in the automated motivational messaging arms were randomized to receive or not receive an automated motivational message). This outcome only applies to participants randomized to receive automated motivational messaging.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-8 (PHQ-8) Self-Report Scale Score - Distal (Long-Term) | 8-week intervention period
  The PHQ-8 is a self-report measure of severity of depressive symptoms. It will be used to determine the impact of the intervention on symptoms of depression.
Change in Generalized Anxiety Disorder-7 (GAD-7) Self-Report Scale Score - Distal (Long-Term) | 8-week intervention period
  The GAD-7 is a self-report measure of severity of anxiety symptoms. It will be used to determine the impact of the intervention on symptoms of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Lipschitz, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Jessica Morrow Lipschitz, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No